CLINICAL TRIAL: NCT01310491
Title: RENEWING HEALTH Large-scale Real-life Study in Finland
Brief Title: RENEWING HEALTH - RegioNs of Europe WorkINg Together for HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Karelia, Social and Health Care District (Other)
Responsible Party: Principal Investigator, Tuula Karhula, Substitute Director of Elderly Services, South Karelia, Social and Health Care District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Renewing Health WP WP 13 Fin
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease; Heart Failure; Atrial Fibrillation; Other Arrhythmias
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usual Care (No Intervention)
  Interventions: Behavioral: Health coaching

INTERVENTIONS:
Behavioral: Health coaching — Telephone based health coaching supported by tele-monitoring.

SUMMARY:
The purpose of this trial is to determine if by structured telephone based health coaching programme supported by remote monitoring system among type 2 diabetes, coronary artery disease and heart failure patients the investigators are able to improve their quality of life as measured by the SF-36 questionnaire and reduce a value of HbA1c under 6,5 % among those type 2 diabetes patients who had elevated value of HbA1c when recruited.

DETAILED DESCRIPTION:
RENEWING HEALTH is a project covering 9 different European States. It aims at evaluation of innovative telemedicine services using a patient-centred approach and a common rigorous assessment methodology. In 9 European regions in the implementation of health-related information and communication technologies service solutions are already operational at local level for the remote monitoring and the treatment of chronic patients suffering from diabetes,chronic obstructive pulmonary disease or cardiovascular diseases. The services are designed to give patients a central role in the management of their own diseases, fine-tuning the choice and dosage of medications, promoting compliance to treatment, and helping health care professionals to detect early signs of worsening in the monitored pathologies. Every area will designed its own real-life trial with certain common elements.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Capability of filling in questionnaires in Finnish language.
* Be able to use Remote Patient Monitoring System
* Be able to use the devices provided
* Has adequate cognitive capacities to participate
* In their medical records, one or both of the following diagnoses:

  a) Type 2 Diabetes, for enrolment
* diagnosed over 3 months prior to the enrolment and
* HbA1c > 6,5 % b) Heart Disease, for enrolment
* Ischemic heart disease or
* Heart Failure or
* Atrial fibrillation or
* Other arrhythmia
* Be able to walk

Exclusion Criteria:

* Not willing to participate (e.g., not willing to sign the consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 12 months
  Health related quality of life is assessed by the SF-36 questionnaire.
HbA1c change over time (participants with T2DM only) | 12 months

SECONDARY OUTCOMES:
Medication compliance | 12 months
Blood pressure reduction | 12 months
Weight reduction | 12 months
Activity increase | 12 months
Smoke cessation | 12 months
Alcohol use reduction | 12 months
Cost for the organization | 12 months
Satisfaction and usability of the technology and equipments. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tuula Karhula, MD, PhD, Principal Investigator — South Karelia social and health district
Locations (1):
- Etelä-Karjalan sosiaali- ja terveydenhuollon kuntayhtymä, Lappeenranta, Finland

REFERENCES:
- [Derived] Karhula T, Vuorinen AL, Raapysjarvi K, Pakanen M, Itkonen P, Tepponen M, Junno UM, Jokinen T, van Gils M, Lahteenmaki J, Kohtamaki K, Saranummi N. Telemonitoring and Mobile Phone-Based Health Coaching Among Finnish Diabetic and Heart Disease Patients: Randomized Controlled Trial. J Med Internet Res. 2015 Jun 17;17(6):e153. doi: 10.2196/jmir.4059. PMID 26084979